CLINICAL TRIAL: NCT06949462
Title: Evaluating the Effectiveness of Large Language Models in Anaesthesia and Procedural Consent: A Comparative Analysis With Traditional Patient Consent Methods
Brief Title: Effectiveness of Large Language Model for Anaesthesia and Procedural Consent
Acronym: PEAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Ke Yuhe, Associate Consultant, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-04-22
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Consent Forms; Anesthesia; Artificial Intelligence (AI)
Keywords: Anaesthesia; Informed Consent; Large Language Model; Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, randomized controlled trial (RCT) design to evaluate the effectiveness of PEAR, a conversational AI chatbot for anaesthesia risk counselling.
  Participants are randomly assigned in a 1:1 allocation ratio to one of two arms:
  Intervention Group: Receives anaesthesia risk information through the PEAR chatbot prior to their consultation with an anaesthetist.
  Control Group: Receives anaesthesia counselling through the standard, face-to-face verbal consent process by a clinician.
  Randomisation is stratified by surgical specialty to ensure balanced representation across different clinical settings.
Who Masked: Outcomes Assessor
Masking Description: There will be no blinding of the participants and investigators due to the impracticality. The outcome assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control arm will receive the standard anaesthesia risk counselling conducted face-to-face by a licensed anaesthetist. This process follows institutional protocols and includes a verbal explanation of anaesthesia procedures, associated risks, benefits, and potential complications, tailored to the patient's specific surgical context.
  Patients are encouraged to ask questions and engage in discussion during the session. No digital tools or chatbot assistance will be used in this arm.
- PEAR (Experimental): Participants in this arm will receive anaesthesia risk counselling through the PEAR (Patient Education of Anaesthesia Risks) chatbot, a multilingual, AI-powered conversational tool. The chatbot provides personalized education on anaesthesia risks, procedures, and post-operative expectations. Patients interact with the chatbot prior to meeting the anaesthetist, enhancing their understanding and preparing them for the face-to-face consultation.
  Interventions: Other: PEAR

INTERVENTIONS:
Other: PEAR — Participants in the intervention arm will receive anaesthesia risk counselling through the PEAR (Patient Education of Anaesthesia Risks) chatbot prior to their face-to-face consultation with an anaesthetist. PEAR is a multilingual, AI-powered conversational tool designed to provide personalized, interactive education on anaesthesia-related procedures, risks, and safety information.
  The chatbot delivers content aligned with institutional guidelines and allows patients to explore topics at their own pace, ask questions in natural language, and revisit information as needed. After completing the chatbot interaction, patients proceed with their standard preoperative consultation, where any further questions are addressed by the anaesthetist.
  This approach is designed to enhance patient understanding, reduce anxiety, and optimize the in-person consultation by preparing patients in advance.
  Arms: PEAR

SUMMARY:
Patient understanding of anaesthesia risks remains inconsistent due to time constraints, language barriers, and variable clinician communication styles. Traditional verbal consent may not consistently ensure comprehension or reduce preoperative anxiety. PEAR (Patient Education of Anesthesia Risks) is a multilingual, AI-driven chatbot developed to enhance patient education and improve the quality of anaesthesia risk counselling.

Study Objective:

To compare PEAR's performance in delivering anaesthesia risk consent against the standard face-to-face verbal method.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of PEAR (Patient Education of Anaesthesia Risks), a conversational AI-based chatbot designed to deliver anaesthesia risk education to patients in a personalized, interactive, and multilingual format. The goal is to support informed consent by improving patient comprehension, satisfaction, and reducing anxiety, while also streamlining clinician workflow.

Participants undergoing elective surgery will be randomly assigned to either receive anaesthesia counselling via PEAR before their consultation with the anaesthetist (intervention group) or undergo the standard face-to-face verbal consent process (control group). The PEAR chatbot is accessed through a secure digital interface and presents information aligned with institutional anaesthesia protocols.

The study will be conducted at hospitals within the SingHealth cluster in Singapore. Following the consent process, patients will complete a short quiz to assess understanding, a survey to evaluate satisfaction, and an anxiety scale. Clinicians will record time taken and perceived workload.

All patients will still meet their anaesthetist, ensuring clinical oversight is maintained. This study does not alter standard care but evaluates a digital adjunct to enhance it. Data will be collected electronically, anonymised, and stored securely. Insights from this trial may inform the wider implementation of digital tools in perioperative patient education.

ELIGIBILITY:
Inclusion Criteria:

- Adults (≥21 years old) undergoing elective surgery requiring anaesthesia

Classified as ASA Physical Status I to III

* Able to provide informed consent
* Able to communicate effectively in English, Chinese (Mandarin), Malay, or Tamil
* Willing and able to complete questionnaires and interact with the PEAR chatbot (intervention arm)

Exclusion Criteria:

* ASA Physical Status IV or above
* Cognitive impairment or psychiatric conditions that may limit comprehension or communication
* Non-literate patients or those unable to understand English, Chinese, Malay, or Tamil
* Emergency surgery cases
* Prior participation in the study (to prevent bias)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient Understanding of Anaesthesia Risks | Immediately post-consent (within 30 minutes of completing the counselling session)
  Patient understanding will be measured using a structured, validated multiple-choice questionnaire immediately after the consent process, specifically the Deaconess Informed Consent Comprehension Test (DICCT). The DICCT evaluates knowledge of key anaesthesia-related risks, safety information, and patient-specific considerations discussed during the counselling session. The DICCT scores range from 0 to 20, with higher scores indicating better understanding and comprehension. This outcome measures the effectiveness of the chatbot (PEAR) compared to traditional verbal consent in conveying critical information and supporting informed decision-making.

SECONDARY OUTCOMES:
Reduction in Patient Anxiety Related to Anaesthesia | Immediately pre-consent and post-consent (within the same clinic visit)
  Patient anxiety levels will be measured using the State-Trait Anxiety Inventory (STAI-S), a validated tool widely used in clinical research. The STAI-S evaluates how anxious a patient feels "right now" (state anxiety) in the context of their upcoming surgery and anaesthesia. The tool includes 20 items rated on a 4-point Likert scale, with higher scores indicating greater anxiety.
  Participants will complete the questionnaire immediately before and after the anaesthesia consent session. Change in anxiety scores will be compared between the intervention (PEAR chatbot) and control (standard verbal consent) groups to evaluate PEAR's effectiveness in reducing preoperative anxiety.
Usability of the PEAR Chatbot Assessed via System Usability Scale (SUS) | Immediately post-chatbot use (same clinic visit)
  Usability of the PEAR chatbot will be assessed using the System Usability Scale (SUS), a validated 10-item questionnaire that measures perceived ease of use, user satisfaction, and learnability of digital tools. Each item is rated on a 5-point Likert scale and results in a score ranging from 0 to 100, with higher scores indicating better usability.
  Patients in the intervention arm (PEAR) will complete the SUS immediately after using the chatbot. This measure will help determine whether the tool is user-friendly and acceptable for perioperative patient education.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the publication (including primary and secondary outcomes, baseline characteristics, and questionnaire scores) will be made available to qualified researchers upon reasonable request.
  Data will be shared beginning 6 months after publication and will be accessible for up to 3 years post-publication. Requests must include a methodologically sound proposal and be submitted to the Principal Investigator. A data access agreement will be required to ensure ethical use and protection of participant confidentiality.
Supporting Information: Analytic Code
Time Frame: 1st July 2025 - 1st july 2028
Access Criteria: Access to de-identified individual participant data (IPD) will be granted to qualified academic researchers, healthcare professionals, or institutions conducting methodologically sound research that aligns with ethical standards and scientific purpose.

REFERENCES:
- [Background] Ke YH, Jin L, Elangovan K, Abdullah HR, Liu N, Sia ATH, Soh CR, Tung JYM, Ong JCL, Kuo CF, Wu SC, Kovacheva VP, Ting DSW. Retrieval augmented generation for 10 large language models and its generalizability in assessing medical fitness. NPJ Digit Med. 2025 Apr 5;8(1):187. doi: 10.1038/s41746-025-01519-z. PMID 40185842